CLINICAL TRIAL: NCT04346173
Title: Palatal Lengthening Using Buccinator Myomucosal Flaps with Furlow Z-plasty Technique for Primary Cleft Palate Repair (A Clinical Study)
Brief Title: Palatal Lengthening Using Buccinator Myomucosal Flaps with Furlow Z-plasty Technique for Primary Cleft Palate Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Akram (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Akram, Assistant lecturer of Oral and Maxillofacial surgery, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Furlow with buccinator
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2020-04

CONDITIONS: Cleft Palate, Unilateral, Complete
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- furlow z plasty with buccinator myomucosal flap (Experimental): using furlow palatoplasty technique accompanied with addition of buccinator myomucosal flap for closure of primary unilateral cleft palate
  Interventions: Procedure: furlow z plasty with buccinator myomucosal flap

INTERVENTIONS:
Procedure: furlow z plasty with buccinator myomucosal flap — using furlow palatoplasty technique accompanied with addition of buccinator myomucosal flap for closure of primary unilateral cleft palate

SUMMARY:
: Cleft palate is a congenital deformity caused by abnormal facial development during intra-uterine life. Worldwide, the prevalence of cleft lip/palate is about 1:1000 live births.

The levator vela palatini muscles are malpositioned sagittally, running postero-anteriorly and inserted onto the posterior edge of the hard palate in cleft palate patients . This configuration prevents the muscle from exerting its upward, backward, and lateral pull.

Various modalities have been described with major refinements over the past 30 years. Gradually, cleft surgeons began to appreciate the importance of dissection and retro-positioning of the levator muscle on improving speech outcomes.

Furlow was the first to describe the palatoplasty technique, in which the levator muscle is dissected and freely released from its abnormal position and retro-positioned in a Z-plasty lengthening technique without dissection on the hard palate. However , among the problems that have been raised concerning the Furlow palatoplasty is the limitation of the procedure in wide clefts. Furthermore, the possibility of higher fistula rate associated with the technique.

These considerations have led to modified palatal lengthening by buccinator myomucosal flaps which is this study working on.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age frame between 9 months and 18 months.
* Cleft palate alone or cleft lip and palate patients.
* Patients who have not done any previous palatal repair
* Haemoglobin level above 10 grams.
* Weight above 10 pounds.

Exclusion Criteria:

* Syndromic patients.
* Medically compromised patients contradicting operation.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
palatal lengthening | immediately postoperative
  measuring the length the palate will gain using this technique

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No